CLINICAL TRIAL: NCT04819568
Title: Comparison of Bolus Versus Continuous Infusion of Terlipressin Cirrhotic Patients With Septic Shock: A Randomized Controlled Trial
Brief Title: Comparison of Bolus Versus Continuous Infusion of Terlipressin Cirrhotic Patients With Septic Shock.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-39
Record Dates: First submitted 2021-03-15; First posted 2021-03-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Terlipressin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terlipressin Bolus Arm (Experimental)
  Interventions: Drug: Terlipressin; Other: Standard of Care
- Terlipressin Continuous Infusion Arm (Active Comparator)
  Interventions: Drug: Terlipressin; Other: Standard of Care

INTERVENTIONS:
Drug: Terlipressin — Terlipressin Bolus Max dose 2 mg/24 hr.i.e 0.5 mg qid
Other: Standard of Care — Standard of Care

SUMMARY:
Septic shock is a major life-threatening vasodilatory shock. Vasopressor form a crucial pharmacotherapeutic option and have long been used as the first and foremost recommended therapy.(1) However, some patients may remain refractory to catecholamine, which is also known as catecholamine-resistant septic shock.(2, 3) High-dose catecholamine therapy may lead to potential side effects such as increased myocardial oxygen consumption, lethal arrthymias, and even the high risk of mortality. (4)Therefore, newer alternatives like dopamine, dobutamine, somatostatin, and terlipressin are also used.

Cirrhosis is a state of hyperdynamic circulation, which worsens with the onset of infection. In septic shock, there is relative deficiency of vasopressin. (13) The mortality of septic shock in these patients still remains extremely high. Terlipressin is a synthetic vasopressin analogue with greater selectivity for the V1-receptors.(5) In cirrhotics with septic shock, terlipressin has been used either as a continuous intravenous infusion or as intravenous boluses. However, at present none of studies reveal which would be a better mode of administration in cirrhotics with septic shock considering the reversal of hemodynamics and safety of patients.

DETAILED DESCRIPTION:
Methodology:

* Study population: All the consecutive patients of cirrhosis admitted to Intensive care unit of Hepatology department of ILBS will be evaluated for inclusion
* Study design: Prospective open label randomised controlled study -superiority trial. The study will be conducted in Department of Hepatology ILBS- intensive care unit.
* Study period: 1 year from ethics approval (Feb 21- Jan 22)
* Sample size: Assuming that the response rate is 90% in continuous and 80% in bolus , with α=5% β=80% and the superiority margin taken as 10%; then we need to enroll 141 cases in each arm, further taking 10% drop out rate, we need to randomise a total of 310 cases (155 in each arm). Randomisation will be done by block randomisation method by taking block size as 10.
* Intervention: 250 patients after screening for all exclusion criteria randomised into 2 arms(group-1, Terlipressin bolus arm) and(group-2, Terlipressin continuous infusion arm) in a ratio 1:1.
* 250 patients after screening for all exclusion criteria randomised into 2 arms(group-1, Terlipressin bolus arm) and(group-2, Terlipressin continuous infusion arm) in a ratio 1:1.
* Monitoring and assessment

Both the group will undergo assessment of cardiac function by measuring NT-Pro BNP, Troponin I, ANP and baseline transthoracic echocardiography (TTE), 30 minutes after the first bolus dose and after the starting of infusion, lastly at 72 hours.

TTE will be performed to evaluate the cardiac function; Cardiac output (velocity time integral at aortic flow times the area of left ventricular outflow tract), LV ejection fraction by modified Simpson's method, LV diastolic function by E/E' measurement, right ventricular systolic function by fractional area change, tricuspid annular plane systolic excursion (TAPSE), and flattening of the interventricular septum.

* USG Doppler will be performed in all the patients to assess the flow in renal, portal, hepatic veins and also permeability index, and extravascular lung volume.
* The macro-hemodynamic parameters were MAP, heart rate, cardiac output, SVR index, global end diastolic volume, extravascular lung water, lung permeability index and hourly urine output. Global tissue perfusion adequacy and microcirculation assessment was done by
* 1. SVR index = MAP-CVP/CO *80 ( 700 - 1500dynes/sec/cm-5
* 2. Global EDV = combined end diastolic volume of all 4 chambers.
* 3. Lactate of Blood Gas preferably
* 4. Lactate clearance13 (defined by lactate baseline-lactate at time point/baseline lactate ×100)
* 5. Central venous O2 saturation (SCV02) with a target of SCVO2>70%
* In all patients, baseline endotoxin activity assay and blood sample will be stored for looking at the effect of therapy on cytokine profile (TNF alpha, IL6, IFN-gamma, and ADAMTS and vWillebrand factor).
* Improvement in Endothelial dysfunction would be assessed by measuring the biomarkers such as Endotoxin, von willebrand factor and ADAMTS at three times At baseline (Hour 0), at 30 minutes after Terlipressin dose and at 72 hours.
* Renal function would be measured by serum Renin, serum cystatin C, urine NGAL,eGFR, and improvement in AKI stage according to KDIGO criteria or requirement of dialysis.
* For assessment of impact of coagulation, ROTEM would be performed at respective time.
* Also the serum level of Noradrenaline and terlipressin will be assessed at starting and after 72 hours.

STATISTICAL ANALYSIS: Continuous data- Student's t test

* Non parametric analysis- Mann Whitney test
* Survival outcome By Kaplan-Meier method curve.
* For all tests, p≤ 0.05 will be considered statistically significant.
* Analysis will be performed using SPSS .
* The analysis will be done with intention to treat and per protocol analysis if applicable.

  - Adverse effects Severity of adverse events (CTACE Grade) GRADE-1
* Loose motion(2 -3 episodes)
* Hyponatremia (135-130) GRADE-2
* Loose motion (4-6 episodes)
* Abdominal pain
* Hyponatremia (130-120) GRADE-3
* Loose motion (> 6)
* Bacterial infections
* Chest pain
* Circulatory overload
* Hponatremia( <120)

GRADE-4

* Arrhythmia
* Myocardial Infarction
* Mesenteric ischemia
* Livedo reticularis
* Respiratory acidosis
* Hepatic encephalopathy
* Gastrointestinal bleeding
* Peripheral cyanosis
* Lactic acidosis
* Bradycardia
* Atrial fibrillation
* Ventricular tachycardia GRADE-5
* Death

  * Stopping Rule: Side effects or toxicities that are severe -arrhythmia, AMI, Cardiomyopathy (defined later) Cyanosis and all orther grade IV adverse effects of Terlipressin.
  * Suspicion or confirmed bowel ischemia.
  * Patient unwilling for further hospital stay.
  * Study unrelated complication here the drug effects could not be assessed (massive GI bleed uncontrolled, bowel perforation or any surgical intervention).

ELIGIBILITY:
Inclusion Criteria:

- Cirrhotics including ACLF with septic shock requiring norepinephrine dose >0.5ug/kg/min to maintain MAP> 65 mm Hg

- An informed consent from the patient or relative

Exclusion Criteria:

* Patients with age less than 18 years or more than 65 years
* Severe known cardiopulmonary disease (Hypertension, structural or valvular heart disease, coronary artery disease, arrhythmias)
* Stroke
* Peripheral Vascular disease
* Gut Paralysis
* Intestinal obstruction
* Cancer, hepato-cellular carcinoma (HCC), intrahepatic or extrahepatic malignancy
* Portal vein thrombosis
* Hepatic vein outflow tract obstruction (HVOTO )
* Pregnancy
* Patients with Pa02/FiO2 ratio <150
* Severe coagulopathy platelets <20,000 and INR > 4
* Active Bleed (Mucosal or variceal)
* Patients already on terlipressin in the last 48 hours
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to give informed consent from family members.
* Patient enrolled in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-03-19 (Estimated); Study Completion 2022-03-19 (Estimated)

PRIMARY OUTCOMES:
Reversal of shock | 72 hours
  DISCONTINUATION OF NOREPINEPHRINE IS CONSIDERED AS REVERSAL OF SHOCK.

SECONDARY OUTCOMES:
Time to reversal of shock | 1 Year
Incidence of adverse effects and discontinuation of therapy due to adverse effects | 24 hours
Incidence of adverse effects and discontinuation of therapy due to adverse effects | Day 3
Impact on AKI (Progression, Resolution, requirement of renal replacement therapy, (RRT) | 24 hours
  AS PER KDIGO STAZE, AKI HAS BEEN DEFINED. INCREMENT OF ONE OR MORE STAZE OR REQUIREMENT OF RRT IS CONSIDERED AS PROGRESSION.
  REMAINING SAME STAZE IS CONSIDERED AS PERSISTENT. DECREMENT OF ONE OR MORE STAZE IS CONSIDERED AS IMPROVEMENT.
Impact on AKI (Progression, Resolution, requirement of renal replacement therapy, (RRT) | Day 3
  AS PER KDIGO STAZE, AKI HAS BEEN DEFINED. INCREMENT OF ONE OR MORE STAZE OR REQUIREMENT OF RRT IS CONSIDERED AS PROGRESSION.
  REMAINING SAME STAZE IS CONSIDERED AS PERSISTENT. DECREMENT OF ONE OR MORE STAZE IS CONSIDERED AS IMPROVEMENT.
Impact on AKI (Progression, Resolution, requirement of renal replacement therapy, (RRT) | Day 7
  AS PER KDIGO STAZE, AKI HAS BEEN DEFINED. INCREMENT OF ONE OR MORE STAZE OR REQUIREMENT OF RRT IS CONSIDERED AS PROGRESSION.
  REMAINING SAME STAZE IS CONSIDERED AS PERSISTENT. DECREMENT OF ONE OR MORE STAZE IS CONSIDERED AS IMPROVEMENT.
Mortality | 28 days
Improvement in SOFA score | 24 hours
  IMPROVEMENT BY ATLEAST 2 POINTS
Improvement in SOFA score | Day 3
  IMPROVEMENT BY ATLEAST 2 POINTS
Lactate clearance | 6 hours
Lactate clearance | 12 hours
  DECREMENT OF 25% LACATATE DELTA LACTATE = CURRENT LACTATE/BASELINE LACTATE *100%
Lactate clearance | 24 hous
  DECREMENT OF 25% LACATATE DELTA LACTATE = CURRENT LACTATE/BASELINE LACTATE *100%
Lactate clearance | 72 hours
  DECREMENT OF 25% LACATATE DELTA LACTATE = CURRENT LACTATE/BASELINE LACTATE *100%
Days of mechanical ventilation | 1 year
Days of Intensive Care Unit stay | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided